CLINICAL TRIAL: NCT01487850
Title: Study of Wind Reed Instruments' Fungal Contamination and Its Immunological and Clinical Consequences for Musicians.
Brief Title: Wind Instruments' Fungal Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Flora METZGER, Medical Doctor, Lung specialist, Principal Investigator, Centre Hospitalier Universitaire de Besancon
Purpose: Diagnostic
Other Study IDs: P/2007/55
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Immunologically-induced Lung Disease; Hypersensitivity Pneumonitis
Keywords: wind instruments; molds; hypersensitivity pneumonitis; fungal contamination of wind instruments; specific antibodies against molds in musicians' sera; musicians
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood sample — blood sample in each musician to search for specific antibodies against molds isolated from instruments

SUMMARY:
On the basis of 2 cases of immunologically-induced lung disease in 2 saxophonists, the investigators supposed that wind reed instruments could be contaminated with molds. The investigators led a study on 40 musicians playing a wind reed instrument to analyze instruments' fungal contamination and its immunological and clinical consequences for musicians.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 year old or more
* must play a wind reed instrument (saxophone, clarinet, bassoon or oboe) one hour per week or more

Exclusion Criteria:

* refuse to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Saint Jacques, Besançon, Franche Comté, France

REFERENCES:
- [Result] Lodha S, Sharma OP. Hypersensitivity pneumonitis in a saxophone player. Chest. 1988 Jun;93(6):1322. doi: 10.1378/chest.93.6.1322. No abstract available. PMID 3371127
- [Result] Metzger F, Haccuria A, Reboux G, Nolard N, Dalphin JC, De Vuyst P. Hypersensitivity pneumonitis due to molds in a saxophone player. Chest. 2010 Sep;138(3):724-6. doi: 10.1378/chest.09-2991. PMID 20822994